CLINICAL TRIAL: NCT07136480
Title: Comparison of the Effectiveness of Various Deep Heating Modalities in the Management of Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Dilara Ekici Zincirci, Medical Doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Low Back Pain
Record Dates: First submitted 2025-08-13; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain
Keywords: low back pain; deep heating modalities; physical therapy
MeSH Terms: conditions — Low Back Pain | interventions — Ultrasonic Therapy

STUDY DESIGN:
Intervention Model Description: This trial was designed as a quasi-experimental, parallel-group study. Participants were allocated to one of the intervention groups in a non-systematic manner, without the use of a formal randomization sequence or allocation concealment. The allocation process aimed to distribute participants evenly across the study arms but did not follow a predefined randomization protocol.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Microwave diathermy + standard lumbar exercise program (Experimental): Continuous mode microwave diathermy (2,450 MHz) will be applied to the lumbar region using a standard physiotherapy unit.
  Interventions: Device: Microwave Diathermy; Behavioral: Lumbar Stabilization and Flexibility Exercise
- Shortwave diathermy + standard lumbar exercise program (Experimental)
  Interventions: Device: Shortwave Diathermy; Behavioral: Lumbar Stabilization and Flexibility Exercise
- Therapeutic ultrasound + standard lumbar exercise program (Experimental)
  Interventions: Device: Therapeutic Ultrasound; Behavioral: Lumbar Stabilization and Flexibility Exercise
- Standard lumbar exercise program only (control) (Active Comparator)
  Interventions: Behavioral: Lumbar Stabilization and Flexibility Exercise

INTERVENTIONS:
Device: Microwave Diathermy — Continuous mode microwave diathermy (2,450 MHz) will be applied to the lumbar region using a standard physiotherapy unit. Each session will last 20 minutes, 5 sessions per week for 3 consecutive weeks, in addition to a standardized lumbar stabilization exercise program.
  Arms: Microwave diathermy + standard lumbar exercise program
Device: Shortwave Diathermy — Continuous mode shortwave diathermy (27.12 MHz) will be delivered to the lumbar region using capacitive or inductive electrodes according to manufacturer guidelines. Each session will last 20 minutes, 5 sessions per week for 3 consecutive weeks, in addition to a standardized lumbar stabilization exercise program.
  Arms: Shortwave diathermy + standard lumbar exercise program
Device: Therapeutic Ultrasound — Continuous mode therapeutic ultrasound at 1 MHz frequency and 1.5 W/cm² intensity will be applied to the lumbar paraspinal muscles with slow circular movements using a coupling gel. Treatment will last 10 minutes per session, 5 sessions per week for 3 consecutive weeks, in addition to a standardized lumbar stabilization exercise program.
  Arms: Therapeutic ultrasound + standard lumbar exercise program
Behavioral: Lumbar Stabilization and Flexibility Exercise — Participants will perform a home-based lumbar stabilization exercise program, including stretching, core strengthening, and posture correction exercises, supervised weekly by a physiotherapist. The program will be performed 3 sessions per week for 4 consecutive weeks.

SUMMARY:
This quasi-experimental, non-randomized, parallel-group clinical trial aims to compare the effectiveness of various deep heating modalities-microwave diathermy, shortwave diathermy, and therapeutic ultrasound-when combined with a standard lumbar exercise program in patients with chronic low back pain. The study will evaluate their effects on pain, functional disability, kinesiophobia, and quality of life. Outcomes will be assessed at baseline and after the 3-week treatment period.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is one of the most prevalent musculoskeletal conditions, often leading to long-term disability, reduced quality of life, and significant socioeconomic burden. Deep heating modalities, such as microwave diathermy, shortwave diathermy, and therapeutic ultrasound, are widely used in physiotherapy practice to reduce pain, improve tissue extensibility, and enhance function. However, direct comparisons of these modalities in CLBP are limited.

This quasi-experimental, non-randomized, parallel-group study will allocate participants to one of four groups:

Microwave diathermy + standard lumbar exercise program

Shortwave diathermy + standard lumbar exercise program

Therapeutic ultrasound + standard lumbar exercise program

Standard lumbar exercise program only (control)

The allocation will be performed in a non-systematic manner without a formal randomization sequence. All participants will receive a standardized home-based lumbar stabilization exercise program, while the intervention groups will also receive their respective deep heating modality in 15 treatment sessions (5/week for 3 weeks).

Primary outcomes will include pain intensity (Visual Analog Scale) and functional disability (Oswestry Disability Index). Secondary outcomes will include kinesiophobia (Tampa Scale for Kinesiophobia) and quality of life (SF-12 PCS and MCS). Assessments will be conducted at baseline and week 3 (post-treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years

Diagnosis of non-specific CLBP >12 weeks

Able to participate in exercise program

Voluntary informed consent provided

Exclusion Criteria:

Specific spinal pathology (tumor, fracture, infection, inflammatory disease)

Lumbar surgery within last 12 months

Pregnancy

Pacemaker or implanted metallic/electronic devices

Neurological deficits

Skin lesions or contraindications to deep heating modalities

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (VAS) | baseline- 3 week
  Pain intensity will be measured using a 100 mm Visual Analog Scale (VAS), where 0 mm represents "no pain" and 100 mm represents "worst imaginable pain
Functional Disability (ODI) | baseline-3 week
  Oswestry Disability Index - ODI: Disability will be evaluated using the ODI (0-100%), where higher percentages indicate greater disability.

SECONDARY OUTCOMES:
Kinesiophobia (Tampa Scale for Kinesiophobia, TSK) | baseline-3 week
  Tampa Scale for Kinesiophobia - TSK:The TSK (17-item version) ranges from 17 to 68 points, with higher scores indicating greater fear of movement/reinjury
Quality of Life (SF-12 PCS & MCS) | baseline-3 week
  Health-Related Quality of Life (Short Form-12 - SF-12 PCS & MCS):The SF-12 provides two component scores: Physical Component Summary (PCS) and Mental Component Summary (MCS). Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşçıoğlu Şehir Hastanesi, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided